CLINICAL TRIAL: NCT00715832
Title: A Phase I Vaccine Study With Autologous Dendritic Cells Loaded With Oncofetal Antigen/iLRP in Patients With Metastatic Breast Cancer
Brief Title: A Phase I Cancer Vaccine Study for Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Cancer Center (Other)
Collaborators: Quantum Immunologics, Inc. (Other); University of South Alabama (Other)
Responsible Party: Paul Schwarzenberger, MD, Quantum Immunologics http://quantumimmunologics.com
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QI-Breast Vaccine 1
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Dendritic cell vaccine; OFA/iLRP; Patients; Line; Chemotherapy; Setting; Four different lines
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Dendritic Cell Vaccination — Autologous dendritic dells will be pulsed with human recombinant oncofetal antigen (OFP/iLRP). The vaccine will be injected intradermally

SUMMARY:
The study uses a molecule or particle that is found only on cancer cells and is unique to cancer cells, as it is not detected on normal tissue. The molecule is known as "oncofetal antigen" or OFA. Because OFA is unique to cancer, the investigators feel OFA could be used to educate the patients' own defenses to more effectively fight the cancer on her own, he or she is harboring. Although investigators found OFA to be present in large concentrations on all cancers, it was found to be especially abundant in breast cancers. Therefore, the investigators feel that this molecule would be a good target for stimulating patient defenses especially against breast cancer cells. To accomplish this, certain defense cells (immune cells) will be washed out from the patients' blood using a machine to which the patient is connected through two small cannulas placed into veins located in the patients' arms. Those cells will be manipulated in the laboratory with artificially engineered OFA. These "reeducated" cells will be injected into the skin of patients. There will be a series of three skin injections in 4 week intervals. It is hoped that this treatment will convert the patients' defenses to a point that effective anti cancer responses will be induced. Effectiveness of the treatment will be monitored with blood tests and assessment of the size of the cancers.

DETAILED DESCRIPTION:
The study is an open-label study to assess safety and immune responses to the universal tumor antigen OFA/iLRP. All patients will be immunized with 1 x 107 viable OFA/iLRP-loaded mature, autologous monocyte-derived dendritic cells (DCs). The DC vaccine will be administered intradermally into the proximal medial upper extremity, contralateral to the original site of breast cancer once every month for 3 months. Changes in the tumor will be documented. The patient will remain in the study unless toxicity or adverse side effects require discontinuation following RECIST and CTC guidelines, or if the patient withdraws for any other reason.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV histologically proven breast cancer as defined by the AJCC Cancer Staging Manual (6 th. Edition 2003).
* Patients must have completed one prior form of chemo and/or radiation therapy for their disease and have failed to achieve remission.
* There must be no clinical or radiographic signs of active brain metastases (CT of brain), or disease to the brain that is not considered controlled.
* At least 4 weeks must have elapsed since chemotherapy or biological therapy and 2 weeks must have elapsed since radiotherapy
* Female patients must be at least 18 years of age
* Must be ambulatory with a ECOG performance status of <2
* Must have common recall antigen DTH skin reaction >2 mm
* Must have lab values as following ANC > 1.5 x 109/L; platelets > 100 x 109/L, Hb> 9 g/dL, creatinine < 1.8 mg/dL or a creatinine clearance > 35 mL/min; total bilirubin < 2 the upper limit of normal, AST and ALT < 2.5 the upper limit of normal; albumin >2.5 g/L
* If of child bearing potential, must practice a reliable method of contraception at screening and must agree to continue this status until 6 months after receiving the last study vaccine injection. An HCG (pregnancy) test will be done monthly until the 3 vaccinations are complete.
* Signed informed consent (see Appendix A, Clinical Protocol section 25.1) to be obtained according to ICH GCP guidelines before the patient is subjected to any extra diagnostic procedures performed for evaluation of eligibility for the trial.

Exclusion Criteria:

* History of other prior malignancy, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or cervical cancer stage IB
* Active infection requiring continuous use of antibiotic therapy
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia
* Autoimmune disease currently treated with steroids
* Adverse reactions to vaccines such as anaphylaxis or other serious reactions, e.g. life-threatening reactions to medicine
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis,systemic lupus erythematosus, scleroderma, polymyositis dermatomyositis, juvenile onset, insulin dependent diabetes, or a vasculitic syndrome
* Pregnancy or lactation
* Any reason why, in the opinion of the investigator, the patient should not participate
* Patients who have received cytotoxic anti-tumor therapy within 4 weeks prior to vaccination
* Patients with active hepatitis (B, C) or HIV+ individuals
* Patients with more than four different lines of chemotherapy in the metastatic setting (excluding adjuvant chemotherapy).

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
toxicity | 24 months

SECONDARY OUTCOMES:
Response, Survival, Immunological Monitoring, Time to Disease Progression | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Quantum Immunologics, Mobile, Alabama, United States

REFERENCES:
- [Background] Holtl L, Zelle-Rieser C, Gander H, Papesh C, Ramoner R, Bartsch G, Rogatsch H, Barsoum AL, Coggin JH Jr, Thurnher M. Immunotherapy of metastatic renal cell carcinoma with tumor lysate-pulsed autologous dendritic cells. Clin Cancer Res. 2002 Nov;8(11):3369-76. PMID 12429623
- [Background] Rohrer JW, Barsoum AL, Dyess DL, Tucker JA, Coggin JH Jr. Human breast carcinoma patients develop clonable oncofetal antigen-specific effector and regulatory T lymphocytes. J Immunol. 1999 Jun 1;162(11):6880-92. PMID 10352310
- [Background] Coggin JH Jr, Barsoum AL, Rohrer JW. 37 kiloDalton oncofetal antigen protein and immature laminin receptor protein are identical, universal T-cell inducing immunogens on primary rodent and human cancers. Anticancer Res. 1999 Nov-Dec;19(6C):5535-42. PMID 10697612
- [Background] Zelle-Rieser C, Barsoum AL, Sallusto F, Ramoner R, Rohrer JW, Holtl L, Bartsch G, Coggin JH JR, Thurnher M. Expression and immunogenicity of oncofetal antigen-immature laminin receptor in human renal cell carcinoma. J Urol. 2001 May;165(5):1705-9. PMID 11342960
- [Background] Coggin JH Jr. Classification of tumor-associated antigens in rodents and humans. Immunol Today. 1994 May;15(5):246-7. doi: 10.1016/0167-5699(94)90251-8. No abstract available. PMID 8024686
- [Background] Barsoum AL, Coggin JH Jr. Isolation and partial characterization of a soluble oncofetal antigen from murine and human amniotic fluids. Int J Cancer. 1991 May 10;48(2):248-52. doi: 10.1002/ijc.2910480216. PMID 1850386
- [Background] Payne WJ Jr, Coggin JH Jr. Mouse monoclonal antibody to embryonic antigen: development, cross-reactivity with rodent and human tumors, and preliminary polypeptide characterization. J Natl Cancer Inst. 1985 Sep;75(3):527-44. PMID 2411994
- [Background] Barsoum AL, Coggin JH Jr. Immunogenicity of a soluble partially purified oncofetal antigen from murine fibrosarcoma in syngeneic mice. J Biol Response Mod. 1989 Dec;8(6):579-92. PMID 2600602
- [Background] Coggin JH Jr, Barsoum AL, Rohrer JW. Tumors express both unique TSTA and crossprotective 44 kDa oncofetal antigen. Immunol Today. 1998 Sep;19(9):405-8. doi: 10.1016/s0167-5699(98)01305-x. No abstract available. PMID 9745203
- [Background] Gussack GS, Rohrer SD, Hester RB, Liu PI, Coggin JH Jr. Human squamous cell carcinoma lines express oncofetal 44-kD polypeptide defined by monoclonal antibody to mouse fetus. Cancer. 1988 Jul 15;62(2):283-90. doi: 10.1002/1097-0142(19880715)62:23.0.co;2-o. PMID 3289728
- [Background] Coggin JH Jr, Rohrer SD, Hester RD, Barsoum AL, Rashid HU, Gussack GS. 44-kd oncofetal transplantation antigen in rodent and human fetal cells. Implications of recrudescence in human and rodent cancers. Arch Otolaryngol Head Neck Surg. 1993 Nov;119(11):1257-66. doi: 10.1001/archotol.1993.01880230105015. PMID 8217085
- [Background] Coggin JH Jr. Oncofetal antigens. Nature. 1986 Jan 30-Feb 5;319(6052):428. doi: 10.1038/319428c0. No abstract available. PMID 3945319
- [Background] Coggin JH Jr, Rohrer JW, Barsoum AL. True immunogenicity of oncofetal antigen/immature laminin receptor protein. Cancer Res. 2004 Jul 1;64(13):4685; author reply 4685. doi: 10.1158/0008-5472.CAN-03-2940. No abstract available. PMID 15231682
- [Background] Rohrer JW, Barsoum AL, Coggin JH Jr. Identification of oncofetal antigen/immature laminin receptor protein epitopes that activate BALB/c mouse OFA/iLRP-specific effector and regulatory T cell clones. J Immunol. 2006 Mar 1;176(5):2844-56. doi: 10.4049/jimmunol.176.5.2844. PMID 16493041
- [Background] Coggin JH Jr. Embryonic antigens in malignancy and pregnancy: common denominators in immune regulation. Ciba Found Symp. 1983;96:28-54. doi: 10.1002/9780470720776.ch3. PMID 6189676
- [Background] Rohrer JW, Culpepper C, Barsoum AL, Coggin JH Jr. Characterization of RFM mouse T lymphocyte anti-oncofetal antigen immunity in apparent tumor-free, long-term survivors of sublethal X-irradiation by limiting dilution T lymphocyte cloning. J Immunol. 1995 Mar 1;154(5):2266-80. PMID 7868899
- [Background] Rohrer JW, Coggin JH Jr. CD8 T cell clones inhibit antitumor T cell function by secreting IL-10. J Immunol. 1995 Dec 15;155(12):5719-27. PMID 7499859